CLINICAL TRIAL: NCT03167710
Title: Electric Dry Needling, Thrust Manipulation and Stretching Versus Impairment-based Manual Therapy, Exercise and Ultrasound for Patients With Lateral Epicondylalgia: A Multi-center Randomized Control Trial
Brief Title: Dry Needling, Manipulation and Stretching vs. Manual Therapy, Exercise and Ultrasound for Lateral Epicondylalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alabama Physical Therapy & Acupuncture (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, James Dunning, DPT, MSc, FAAOMPT, Primary Investigator and President of Spinal Manipulation Institute and Dry Needling Institute of the American Academy of Manipulative Therapy, Alabama Physical Therapy & Acupuncture
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAMT0010
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Dry Needling; Musculoskeletal Manipulations; Exercise; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dry needling, manipulation stretching (Experimental)
  Interventions: Other: Dry Needling, manipulation, stretching
- manual therapy, exercise, ultrasound (Active Comparator)
  Interventions: Other: manual therapy, exercise, ultrasound

INTERVENTIONS:
Other: Dry Needling, manipulation, stretching — HVLA thrust manipulation to elbow, wrist and spine (C5-C6). Dry needling to wrist extensor muscles on the dorsal forearm, proximal and distal of the lateral epicondyle. Up to 8 treatment sessions over 4 weeks.
  Arms: dry needling, manipulation stretching
Other: manual therapy, exercise, ultrasound — Impairment-based manual therapy, exercise and ultrasound targeting the wrist extensors on the dorsal forearm, proximal and distal of the lateral epicondyle. Up to 8 treatment sessions over 4 weeks.
  Arms: manual therapy, exercise, ultrasound

SUMMARY:
The purpose of this research is to compare two different approaches for treating patients with lateral epicondylalgia: electric dry needling, thrust manipulation and stretching versus impairment-based manual therapy, exercise and ultrasound. Physical therapists commonly use all of these techniques to treat lateral epicondyalgia. This study is attempting to find out if one treatment strategy is more effective than the other.

DETAILED DESCRIPTION:
Patients with epicondyalgia will be randomized to receive 2 treatment sessions per week for 4 weeks (up to 8 sessions total) of either: (1) electric dry needling, thrust manipulation and stretching or (2) impairment-based manual therapy, exercise and ultrasound

ELIGIBILITY:
Inclusion Criteria:

1. Adult between 18 and 60 years old that is able to speak English.
2. Report of at least 6 weeks of elbow (i.e. lateral epicondyle) and dorsal forearm pain, consistent with lateral epicondylitis:
3. Patient has not had physical therapy, massage therapy, chiropractic treatment or injections for elbow pain in the last 6 months:
4. Diagnosis of lateral epicondylitis, defined as two of more of the following:

   1. Pain on palpation over the lateral epicondyle and the associated common extensor unit
   2. Pain on gripping a hand dynamometer
   3. Pain with stretching or contraction of the wrist extensor muscles

Exclusion Criteria:

1. Report of red flags to manual physical therapy to include: severe hypertension, infection, uncontrolled diabetes, peripheral neuropathy, heart disease, stroke, chronic ischemia, edema, severe varicosities, tumor, metabolic disease, prolonged steroid use, fracture, RA, osteoporosis, severe vascular disease, malignancy, etc.
2. Report of Previous surgery of the elbow, history of elbow dislocation, elbow fracture and/or tendon rupture
3. Report of systemic neurological disorders and/or neurological deficits to include the following:

   1. Nerve root compression (muscle weakness involving a major muscle group of the upper extremity, diminished upper extremity deep tendon reflex, or diminished or absent sensation to pinprick in any upper extremity dermatome)
   2. Cervical spinal stenosis (exhibited bilateral upper extremity symptoms)
   3. Central nervous system involvement (hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes)
   4. History of whiplash injury within the previous 6 weeks
4. History of surgery to the head/neck or affected upper extremity.
5. Psychiatric disorders or cognitively impaired
6. Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Elbow pain (NPRS) (Rating Score) | Baseline, 1 week, 4 weeks, 3 months
  Rating Score. Baseline score must exceed 2/10 to be included in the study.
Change in Patient-related Tennis Elbow Questionnaire | Baseline, 1 week, 4 weeks, 3 months
  The pain, disability-specific activities and disability common activities section of the PRTEE are collectively measured on a 0-150 point scale. Greater scores indicate increased disability. Baseline must exceed 10/50 on the pain section, 10/60 on the specific activities section and 10/40 on the common activities to be included in the study.

SECONDARY OUTCOMES:
Change in Global Rating of Change Score | 1 week, 4 weeks, 3 months
Change in Tennis Elbow Functional Scale | Baseline, 1 week, 4 weeks, 3 months
  The Tennis Elbow Functional Scale (TEFS) is a 0-40 that assesses disability related to lateral epicondylitis. Greater scores indicate increased disability.
Change in Medication Intake (Frequency of medication intake in last week) | Baseline, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: James Dunning, DPT, Principal Investigator — American Academy of Manipulative Therapy
Locations (1):
- Evolution Sports Physiotherapy, Cockeysville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Young I, Dunning J, Mourad F, Escaloni J, Bliton P, Fernandez-de-Las-Penas C. Clinimetric analysis of the numeric pain rating scale, patient-rated tennis elbow evaluation, and tennis elbow function scale in patients with lateral elbow tendinopathy. Physiother Theory Pract. 2025 Aug;41(8):1712-1720. doi: 10.1080/09593985.2025.2450090. Epub 2025 Jan 10. PMID 39793982
- [Derived] Dunning J, Mourad F, Bliton P, Charlebois C, Gorby P, Zacharko N, Layson B, Maselli F, Young I, Fernandez-de-Las-Penas C. Percutaneous tendon dry needling and thrust manipulation as an adjunct to multimodal physical therapy in patients with lateral elbow tendinopathy: A multicenter randomized clinical trial. Clin Rehabil. 2024 Aug;38(8):1063-1079. doi: 10.1177/02692155241249968. Epub 2024 Apr 26. PMID 38676324